CLINICAL TRIAL: NCT03493373
Title: Effect of Nervous System Mobilization on Older Adults' Postural Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/2018
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Older Adults
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and nervous system mobilization (Experimental): This group will receive neural mobilization and therapeutic exercise: two sessions of 60 minutes during 8 weeks.
  Interventions: Other: Exercise; Other: Neural mobilization
- Exercise (Experimental): This group will receive therapeutic exercise: two sessions of 60 minutes during 8 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The exercise program will consist of: 1) warm up - consisting of stretches of large muscle groups of the upper limbs, lower limbs and trunk and by general mobility exercises; 2) strength training of moderate intensity; 3) balance training; 4) Cooling - will consist of performing overall stretching combined with deep breathing.
Other: Neural mobilization — Neural gliding mobilization will target mainly the lower limb nerves and will be performed in series of 10 repetitions with 1 minute interval between series.
  Arms: Exercise and nervous system mobilization

SUMMARY:
This study aims to compare the effectiveness of nervous system mobilization and exercise with exercise only on institutionalized older adults' postural control.

DETAILED DESCRIPTION:
It is anticipated that 26 institutionalized older adults will be randomly allocated to receive either exercise and neural mobilization (n=13) or exercise only (n=13).

Data on pain intensity (a vertical numeric rating scale) and location (body chart), depression (Geriatric Depression Scale), balance, hand grip strength, timed up and go and gait velocity will be collected at baseline, end of treatment and at 3 months follow up.

Statistical analysis will be performed using a mixed-methods ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* be 65 years of age or older;
* to have independent gait with or without technical aid;
* have indication of the institution's doctor for participation in the study

Exclusion Criteria:

* inability to understand study aims.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Gait velocity | Baseline
  Participants are asked to walk at normal gait velocity over 4 meters and gait velocity is calculated
Gait velocity | 9 weeks
  Participants are asked to walk at normal gait velocity over 4 meters and gait velocity is calculated
Gait velocity | 3 months
  Participants are asked to walk at normal gait velocity over 4 meters and gait velocity is calculated

SECONDARY OUTCOMES:
Pain intensity | Baseline
  Pain intensity measured using a vertical numeric rating scale (Range: 0 to 10 and higher values are indicative of higher pain intensity)
Pain intensity | 9 weeks
  Pain intensity measured using a vertical numeric rating scale (Range: 0 to 10 and higher values are indicative of higher pain intensity)
Pain intensity | 3 months
  Pain intensity measured using a vertical numeric rating scale (Range: 0 to 10 and higher values are indicative of higher pain intensity)
Pain location | Baseline
  Measured using a body chart (a graphic representation of the body) where participants identify painful body sites
Pain location | 9 weeks
  Measured using a body chart (a graphic representation of the body) where participants identify painful body sites
Pain location | 3 months
  Measured using a body chart (a graphic representation of the body) where participants identify painful body sites
Depressive symptoms | Baseline
  Measured using the 15-itens Geriatric Depression Scale (range: 0-15; participants who score 5 or more have depression)
Depressive symptoms | 9 weeks
  Measured using the 15-itens Geriatric Depression Scale (range: 0-15; participants who score 5 or more have depression)
Depressive symptoms | 3 months
  Measured using the 15-itens Geriatric Depression Scale (range: 0-15; participants who score 5 or more have depression)
Balance | Baseline
  Participants are asked to maintain a tandem/semi-tandem position for up to 30 seconds.
Balance | 9 weeks
  Participants are asked to maintain a tandem/semi-tandem position for up to 30 seconds.
Balance | 3 months
  Participants are asked to maintain a tandem/semi-tandem position for up to 30 seconds.
Timed up and go test | Baseline
  Get up from a chair, walk 3 meters, go back to the chair and sit back. The amount of time that each participant takes to perform the task is taken.
Timed up and go test | 9 weeks
  Get up from a chair, walk 3 meters, go back to the chair and sit back.The amount of time that each participant takes to perform the task is taken.
Timed up and go test | 3 months
  Get up from a chair, walk 3 meters, go back to the chair and sit back. The amount of time that each participant takes to perform the task is taken.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Lar Santa Catarina do Reboleiro, Guarda
  - Lar da Santa Cruz da Beselga, Guarda

IPD SHARING:
Plan to Share IPD: No